CLINICAL TRIAL: NCT03417804
Title: Incidence of Postoperative Residual Neuromuscular Blockade - A Multicenter, Observational Study in Portugal
Brief Title: Incidence of Postoperative Residual Neuromuscular Blockade in Portugal
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Simao Esteves, MD, Centro Hospitalar do Porto
Other Study IDs: 2017.156(133-DEFI/125-CES)
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Residual Neuromuscular Blockade; Residual Paralysis, Post-Anesthesia; Observational Study; Complication of Anesthesia; Neuromuscular Blockade
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an epidemiological multicenter, observational, prospective study, designed to determine the incidence of postoperative residual neuromuscular blockade - defined by a TOF (train-of-four) ratio < 0.9 - at PACU arrival.

Subjects aged at least 18 years old (n=360) admitted for different types of elective surgical procedures requiring general anesthesia with neuromuscular blocking agents will be included.

DETAILED DESCRIPTION:
This is a multicenter, observational/non-interventional study involving adult patients undergoing different types of elective surgical procedures requiring general anesthesia with neuromuscular blocking agents.

The study will have two periods:

* Period 1 - Evaluation at PACU arrival.
* Period 2 - Collection of hospital patient discharge data.

A total of 360 patients will be included from approximately 10 centers in Portugal, where the PACU is adjacent to the Operating Room (OR). Each center should recruit between 30 and 40 patients.

Each subject is considered to be enrolled in the study when the subject has provided written informed consent.

Enrollment will be stopped when approximately 360 patients are recruited.

A subject is considered to have completed the trial after all of the protocol specified activities are completed. A subject is considered to have discontinued after he/she has withdrawn consent or has been discontinued.

Overall, study start is when the first site is initiated and study ends at database lock.

During the routine preoperative anesthesia visit the patient will be asked to participate in the study. A description of the study will be provided to the patient by the investigator or qualified designee and any questions will be properly answered. If the patient agrees to participate in the study an informed consent form (ICF) will be signed.

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion. A copy of the signed and dated consent form should be given to the subject before participation in the study.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/ERC's (Institutional Review Board) ) approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the study.

All consented subjects will be given a unique patient number that will be used to identify the subject for all procedures. Each subject will be assigned only one patient number.

Immediately after patient arrival in the PACU and as soon as clinically adequate (basic monitoring and oxygen therapy in place) the anesthesiologist assigned to the PACU (who was not involved in the anesthetic procedure) will collect demographic data (gender, age, weight, height), vital signs (heart rate, blood pressure, oxygen saturation and temperature). Neuromuscular blockade (TOF Ratio) will be measured. Clinical history, co-morbidities, surgical diagnosis, ASA (American Society of Anesthesiology) classification and perioperative medication data (dosage and last administration time) will be collected as well.

As this is an observational study, intra-operative monitoring of neuromuscular blockade will not be mandatory by protocol and will be left at the discretion of the anesthesiologist as according to the clinical practice. Only information about whether this evaluation was performed or not, and if yes if it was used quantitative or qualitative methods, will be collected in the CRF (case report form) .

Neuromuscular blockade evaluation Neuromuscular blockade will be evaluated using a quantitative method. Three consecutive TOF stimulations will be applied. In case these 3 measures differ more than 20%, another sequence of 3 consecutive TOF measurements will be considered. If after the 2nd sequence the 3 consecutive TOF measurements still differ more than 20% between the maximum and the minimum the patient will be excluded.

This study will reflect real life clinical practice. The anesthetic technique in terms of drugs and type of monitoring used will be of entire responsibility of the anesthesiologist.

All study activities will be consistent with EU (European Union) directive 2001/20/EC section for non- interventional studies :

* NMBAs (neuromuscular blocking agents) and reversal agents (as well as all drugs which will be used during the anesthesia) administration will be done in accordance with routine anesthesiology practice and labeling of these medicine products;
* No further interventional means, methods or procedures, are scheduled for subjects, which would otherwise not be applied;
* Furthermore, there will be no additional visits to the hospital or a mandatory visit schedule, deviating from daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Informed consent signed;
* Admission for elective surgery;
* Administration of non-depolarizing NMBAs during surgery

Exclusion Criteria:

* Admission for emergency surgery;
* Reoperation on the same hospital admission;
* More than 10 minutes elapsed between extubation and neuromuscular block monitoring at PACU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery on 10 centers that accepted to participate in the study.
Sampling Method: Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simao Esteves, MD, Principal Investigator — Centro Hospitalar do Porto
Locations (10):
- Portugal (10):
  - Hospital Prof. Fernando Fonseca, EPE, Amadora
  - Centro Hospitalar Baixo Vouga, Aveiro
  - Centro Hospitalar Universitário de Coimbra, Coimbra
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Centro Hospitalar Tamega Sousa, Penafiel
  - Centro Hospitalar do Porto, Porto
  - Centro Hospitalar S. João, Porto
  - Centro Hospitalar Vila Nova Gaia/Espinho, Vila Nova de Gaia
  - Centro Hospitalar Tondela Viseu, Viseu

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients > 18 years old submitted to surgery under general anesthesia with the use of non-depolarizing neuromuscular blocking agents from 10 public Portuguese hospitals
Groups:
- Patients Proposed for Elective Surgical Procedures: A multicentre prospective observational study in adult patients undergoing different types of elective surgical procedures requiring general anaesthesia with non-depolarizing NMBAs was conducted between July 2018 and July 2019 at 10 public Portuguese hospitals
Period: Overall Study
Arm/Group | Patients Proposed for Elective Surgical Procedures
Started | 366 (at least 360 patients)
Completed | 366
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Proposed for Elective Surgical Procedures
Number analyzed (Participants) | 366
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [48 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207
  Male | 159
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Portugal | 366

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Postoperative Residual Neuromuscular Blockade
Description: Percentage of patients arriving PACU with a TOF ratio < 0.9 measured as average of 3 consecutive TOF stimulations
Time Frame: No more than 10 minutes after operating room exit
Measure: Count of Participants; unit: Participants
Groups:
- Patients Proposed for Elective Surgical Procedures: A multicentre prospective observational study in adult patients undergoing different types of elective surgical procedures requiring general anaesthesia with non-depolarizing NMBAs was conducted between July 2018 and July 2019 at 10 public Portuguese hospitals
  20 patients out of 366 presented with TOFr< 0.9 which represents an incidence of 5,5%
Arm/Group | Patients Proposed for Elective Surgical Procedures
Number analyzed (Participants) | 366
Participants | 20

2. Secondary Outcome: Percentage of Patients With Severe Residual Postoperative Neuromuscular Blockade
Description: Percentage of patients with severe postoperative residual neuromuscular blockade defined by a TOF ratio < 0.7
Time Frame: no more than 10 minutes after operating room exit
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Proposed for Elective Surgical Procedures
Number analyzed (Participants) | 366
Participants | 2

3. Secondary Outcome: Association of Postoperative Residual Blockade and the Use of Reversal Agents
Description: Association of postoperative residual blockade and the use of reversal agents (neostigmine, sugammadex or none)
Time Frame: no more than 10 minutes after operating room exit
Reporting Status: Not Posted

4. Secondary Outcome: Association of Postoperative Residual Blockade and the Use of Intra-operative Monitoring of Neuromuscular Blockade
Description: To evaluate the association of postoperative residual blockade and the use of intra-operative monitoring of neuromuscular blockade
Time Frame: no more than 10 minutes after operating room exit
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Association of Postoperative Residual Blockade and ASA Status
Description: To evaluate the association of postoperative residual blockade with co- morbidities and ASA status
Time Frame: no more than 10 minutes after operating room exit
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 day
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Arm/Group | Patients Proposed for Elective Surgical Procedures
All-Cause Mortality (participants affected / at risk) | 0/366
Serious Adverse Events (participants affected / at risk) | 2/366
Other Adverse Events (participants affected / at risk) | 10/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Proposed for Elective Surgical Procedures (N=366)
Pulmunary thromboembolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Severe residual neuromuscular blockade (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Proposed for Elective Surgical Procedures (N=366)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Sore throat (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to its observational nature, it was not possible to standardize practices between centres.

A convenience sample was used (patients were included when investigators were scheduled to PACU), what may have biased the study sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT03417804/Prot_SAP_001.pdf